CLINICAL TRIAL: NCT00202839
Title: Comparison of the Sustained Response of Peg-Intron/Ribavirin Combination Therapy in Genotype 1-Infected Hepatitis C Patients for Non-extended Versus 24-week Extended Treatment After 24 Weeks Pilot Treatment in Taiwan
Brief Title: Peg-Intron/Ribavirin in G 1 HCV for Non-Extended Versus 24 Week Extended Treatment After 24 Weeks (Study P04144)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04144
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24-Week Treatment (Experimental): Genotype 1 hepatitis C virus [HCV] subjects treated for a total of 24 weeks, during the pilot treatment program (immediately before randomization)
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Ribavirin
- 48-Week Treatment (Active Comparator): Genotype 1 HCV subjects treated for a total of 48 weeks: 24 weeks during the pilot treatment program (immediately before randomization) plus 24 weeks during the extended treatment program (immediately after randomization)
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Ribavirin

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — Powder for injection in vial (120 microgram strength), subcutaneous, dose of 1.5 micrograms/kg weekly for 24 weeks during the pilot treatment program
  Other Names: peginterferon alfa-2b; SCH 54031
  Arms: 24-Week Treatment
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — Powder for injection in vial (120 microgram strength), subcutaneous, dose of 1.5 micrograms/kg weekly for 24 weeks during the pilot treatment program followed by 1.2 to 1.5 microgram/kg weekly for 24 weeks during the extended treatment program
  Other Names: peginterferon alfa-2b; SCH 54031
  Arms: 48-Week Treatment
Drug: Ribavirin — 200 mg capsules, oral, weight-based dose of 1000 or 1200 mg, daily for for 24 weeks during the pilot treatment program
  Other Names: SCH 18908
  Arms: 24-Week Treatment
Drug: Ribavirin — 200 mg capsules, oral, weight-based dose of 1000 or 1200 mg, daily for for 24 weeks during the pilot treatment program and for 24 weeks during the extended treatment program
  Other Names: SCH 18908
  Arms: 48-Week Treatment

SUMMARY:
This is an open-label, randomized, comparative, multicenter, 48-week study designed to evaluate the efficacy and safety of combination treatment with pegylated interferon and ribavirin in adult subjects with a diagnosis of compensated chronic hepatitis C (hepatitis C virus (HCV)-ribonucleic acid (RNA) positive) (Genotype 1). All subjects will complete 24 weeks of treatment, termed the Pilot Treatment Program, after which all eligible subjects will be randomly assigned to one of two study groups. One group will be followed for an additional 48 weeks without study medication, while the other will be continuously treated for an additional 24 weeks and then followed for another 24 weeks without study medication. Sustained virologic response, defined as undetectable HCV-RNA in serum at the end of the follow-up period, will be measured along with other outcomes.

DETAILED DESCRIPTION:
This is an open-label, randomized, comparative, multicenter study for evaluation of PegIntron/Ribavirin therapy in the efficacy and safety in adult subjects with a diagnosis of compensated chronic hepatitis C (HCV-RNA+) (Genotype 1). This is a 48-week study, for which all subjects should participate in the Pilot Treatment Program and complete 24 weeks treatment. To avoid a treatment gap, subjects who will be screened and eligible subjects will sign informed consent prior to the end of the Pilot Treatment Program. After completion of the Pilot Treatment Program, all eligible subjects will be randomly assigned to either study group. Subjects in the 24-Week Treatment arm will be followed-up without study medication for 48 weeks; subjects in the 48-Week Treatment arm will be continuously treated for another 24 weeks and all subjects in the 48-Week Treatment arm will be followed for another 24 weeks after completion of the treatment period. Subjects in both arms will be evaluated at screening, randomization, 4, 8, 12, 16, 20, 24, 28, 36 and 48 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Males and non-pregnant females and aged >= 18 years, subjects who are over 65 years of age must be in generally good health and must be discussed with and approved by the principal investigator prior to entry.
* The laboratory evaluation within 6 months prior to entering the Pilot Treatment Program must meet the following criteria:
* Hemoglobin values of >= 12 g/dL for females and >= 13 g/dL for males
* Neutrophil count >= 1.5 X10^9/L
* Platelets count >= 100 x 10^9/L
* Total bilirubin < 1.5 mg/dL
* Serum creatinine within normal limits
* Positive serum HCV-RNA (>= 50 IU (100 copy numbers)/mL)
* Anti-HCV positive
* Available HCV genotype 1
* Liver biopsy performed within 12 months prior to entry to this protocol with a pathology report confirming that the histological diagnosis is consistent with chronic hepatitis (METAVIR system >=F1).
* Compensated liver disease with the following hematological, biochemical, and serologic criteria at the screening visit:
* Hemoglobin values of >= 9 g/dL
* Neutrophil count >= 0.75 x 10^9/L
* Platelets count >= 50 x 10^9/L
* Prothrombin time (PT) prolong <= 3 sec, International Normalized Ratio (INR) <= 1.2
* Total bilirubin <= 3 mg/dL
* Within normal limits (subjects requiring medication to maintain TSH levels in the normal range are eligible if all other inclusion/exclusion criteria are met).
* Anti-Human Immunodeficiency Virus (HIV) negative.
* Alpha-fetoprotein (AFP) value within normal limits obtained within 12 months prior to entry. Results above the upper limit of normal but <= 50 ng/mL require both of the following:
* AFP value <= 50 ng/mL obtained within 9 months prior to entry in the study or during the Screening period, and Ultrasound obtained within 9 months prior to entry or in the screening period in the study for evidence of not having hepatocellular carcinoma.
* A urine pregnancy test obtained prior to the initiation of pilot treatment must be negative. Female subjects must not be breast feeding.
* Reconfirmation that sexually-active subjects are practicing acceptable methods of contraception during screening period.
* Complete 24 weeks treatment of the Pilot Treatment Program with Peg-Intron + Ribavirin.
* Must be never treated with interferon for HCV infected hepatitis (treatment naïve) before the Pilot Treatment Program.
* The total amount of Peg-Intron and Ribavirin received during the pilot treatment program must achieve more than 80% of the recommended dosage.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Have decompensated cirrhosis.
* History of severe psychiatric disease, especially depression.
* Concurrent malignancies (including hepatocellular carcinoma).
* Unstable or significant cardiovascular diseases. Subjects with (ECG) showing clinically significant abnormalities.
* Prolonged exposure to known hepatotoxins such as alcohol or drugs.
* History of thyroid disease poorly controlled on prescribed medication.
* Poorly controlled diabetes mellitus.
* Has suspected or confirmed significant hepatic disease from an etiology other than HCV.
* Patients co-infected with hepatitis B and /or human immunodeficiency virus (HIV).
* Severe renal disease or myeloid dysfunction.
* History of organ transplantation other than cornea and hair transplant.
* Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.
* Any other condition which in the opinion of the investigator would make the subject unsuitable for enrollment, or could interfere with the subject participating in and completing the protocol.
* Allergy to interferon.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Shinn Chen, MD, Study Chair — Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 24-Week Treatment | 48-Week Treatment
Started | 78 | 82
Completed | 54 | 72
Not Completed | 24 | 10
Not completed — Adverse Event | 1 | 5
Not completed — Physician Decision | 12 | 0
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24-Week Treatment | 48-Week Treatment | Total
Number analyzed (Participants) | 78 | 82 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.63 (10.6) | 50.46 (10.93) | 50.55 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 39 | 59
  Male | 58 | 43 | 101
Region of Enrollment [Number; unit: participants]
  Taiwan, Province Of China | 78 | 82 | 160

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Achieved a Sustained Virologic Response (SVR)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid [HCV-RNA] levels below assay detection 24 weeks after termination of anti-HCV therapy
Time Frame: 24 weeks of follow-up after either 24 or 48 weeks of anti-HCV therapy
Population: Intention to treat [ITT] population defined as participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | 24-Week Treatment | 48-Week Treatment
Number analyzed (Participants) | 78 | 82
Percentage of participants | 56.41 | 67.07
Statistical Analysis 1: Comparison: 24-Week Treatment vs 48-Week Treatment; Test type: Superiority or Other; p = 0.1651, Chi-squared

2. Secondary Outcome: The Percentage of Participants Who Achieved a Virologic Response 48 Weeks After Randomization.
Description: Virologic response was defined as undetectable HCV-RNA level in the blood.
Time Frame: 48 weeks after randomization (with 24 weeks of treatment immediately before randomization and either 0 or 24 weeks of treatment immediately after randomization)
Population: Intention to treat [ITT] population
Measure: Number; unit: Percentage of Participants
Arm/Group | 24-Week Treatment | 48-Week Treatment
Number analyzed (Participants) | 78 | 82
Percentage of Participants | 57.69 | 67.07

ADVERSE EVENTS:
Arm/Group | 24-Week Treatment | 48-Week Treatment
Serious Adverse Events (participants affected / at risk) | 5/78 | 8/82
Other Adverse Events (participants affected / at risk) | 29/78 | 47/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24-Week Treatment (N=78) | 48-Week Treatment (N=82)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOCAL SWELLING (General disorders) | 0 (0) | 1 (1)
NODULE (General disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 2 (2)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BLOOD GLUCOSE ABNORMAL (Investigations) | 1 (1) | 0 (0)
SEVERE THROMBOCYTOPENIA (Investigations) | 0 (0) | 1 (1)
FISTULA DISCHARGE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24-Week Treatment (N=78) | 48-Week Treatment (N=82)
THYROID DISORDER (Endocrine disorders) | 2 (3) | 5 (8)
FATIGUE (General disorders) | 4 (4) | 5 (7)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 8 (9)
MALAISE (General disorders) | 3 (3) | 5 (7)
PYREXIA (General disorders) | 0 (0) | 8 (11)
NASOPHARYNGITIS (Infections and infestations) | 4 (5) | 2 (2)
ALANINE AMINOTRANSFERASE ABNORMAL (Investigations) | 5 (8) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (5) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (5) | 1 (1)
HAEMOGLOBIN ABNORMAL (Investigations) | 0 (0) | 9 (9)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
HEADACHE (Nervous system disorders) | 3 (3) | 6 (7)
INSOMNIA (Psychiatric disorders) | 8 (8) | 11 (16)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (10)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator and Institution further agree to provide forty-five (45) days written notice to Sponsor prior to submission for publication or presentation to permit Sponsor to review drafts of abstracts and manuscripts for publication.